CLINICAL TRIAL: NCT04950868
Title: A Pilot Study on the Safety, Tolerability, and Effectiveness of Quetiapine in Postpartum Depression
Brief Title: The Safety, Tolerability, and Effectiveness of Quetiapine in Postpartum Depression
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Verinder Sharma (Other)
Responsible Party: Sponsor-Investigator, Verinder Sharma, Principal investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 118885
Record Dates: First submitted 2021-06-11; First posted 2021-07-06 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Postpartum Depression
Keywords: Quetiapine; postpartum; Drug therapy; Major depressive disorder
MeSH Terms: conditions — Depression, Postpartum; Depressive Disorder, Major | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quetiapine (Experimental): They will initially be given 25 mg of quetiapine per day. The dose may be increased by 25-50 mg per week, to a maximum dose of 150 mg per day by week 6 of the study.
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Quetiapine — They will initially be given 25 mg of quetiapine per day. The dose may be increased by 25-50 mg per week, to a maximum dose of 150 mg per day by week 6 of the study.

SUMMARY:
Postpartum depression is a serious disorder that affects approximately 14% of women who have recently given birth. Postpartum depression is either an episode of major depressive disorder (only low periods) or bipolar disorder (periods of lows and highs).

Untreated postpartum depression can negatively affect the mother, the infant and the family. Antidepressants are the most used treatments; however, for many women these drugs are not useful, resulting in a pressing need for effective treatments for postpartum depression. Lack of sleep is common after delivery and can trigger depression in some women. Quetiapine, a drug used for bipolar disorder, major depressive disorder and occasionally sleeplessness has not been well studied in postpartum depression. This study aims to find out how mothers tolerate the drug and whether it is effective for postpartum depression. Results of this study may help investigators carry out a larger study comparing quetiapine and placebo (a sugar pill) in postpartum depression.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient woman between ages 18 - 45
* Within 6 months of delivery
* Have a DSM-5 diagnosis of MDD or BD I, BD II or other specified bipolar or related disorder with peripartum onset
* Have a score of >18 on the 17-item Hamilton Depression Rating Scale (HDRS)
* Have a score of ≤12 Young Mania Rating Scale (YMRS) at both the screening and baseline visits
* Able to communicate in English
* Capable of providing informed consent

Exclusion Criteria:

* A diagnosis of schizophrenia spectrum or other psychotic disorders, obsessive-compulsive disorder, eating disorders, substance-related and addictive disorders
* At high risk for suicide (actively suicidal or a score of ≥ 3 on item #3 on the HDRS)
* Receiving a psychotropic drug such a mood stabilizer, an antidepressant or a sedative/hypnotic.
* Receiving psychotherapy
* Have a physical illness that is a contraindication to the use of quetiapine, or who have a history of intolerance or nonresponse to quetiapine
* Pregnant or planning on becoming pregnant during the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment and retention rate | 10 weeks
  Data on the recruitment rate, refusal rate, retention rate will be used to assess feasibility
Blood pressure | 8 weeks
  The measurement of blood pressure (both systolic and diastolic blood pressure) will be measured in mm HG
Incidence of Treatment-Emergent Adverse Events as assessed by the Systematic Monitoring of Adverse events Related to TreatmentS (SMARTS) score | 8 weeks
  The Systematic Monitoring of Adverse events Related to TreatmentS (SMARTS), will be used to gather information about side effects of quetiapine. It is a check list to identify potential side effects.
Maternal functioning will be measured by the Barkin Index of Maternal Functioning (BIMF) | 8 weeks
  Tolerability described as the degree to which overt adverse effects are tolerated, will be measured using the Barkin Index of Maternal Functioning (BIMF). The Barkin Index of Maternal Functioning score from baseline to week 8 will also be assessed. The sum of the scores is calculated, ranging from 0 to 120. Where a score of 120 means perfect functioning. The different between the scores scores will be looked at and a more positive score (8 week score is greater than baseline score) is a better outcome.
Pulse | 8 weeks
  Pulse will be measured in beats per minute
Body mass index | 8 weeks
  Weight (km) and height (m) will be used to calculate BMI (kg/m^2)
Fasting lipid panel test | 8 weeks
  The fasting lipid panel will be completed to measure safety of the intervention. This measures lipid levels (Total Cholesterol, High Density Lipoprotein, Low Density Lipoprotein, and Triglycerides). All measured in mg/dL
glycated haemoglobin (HbA1c) tests | 8 weeks
  Glycated haemoglobin (HbA1C) test will be done to measure glycated haemoglobin which will measure the safety of the intervention. It will be measured in mmol/mol and as a percentage.
Waist circumference | 8 weeks
  Waist circumference (cm) will help measure the safety of the intervention
Returned tablet count | 8 weeks
  Adherence will be determined by returned tablet count.

SECONDARY OUTCOMES:
Hamilton Depression Rating (HDRS) total score | 8 weeks
  Secondary outcome will be the mean change from baseline to week 8 in the Hamilton Depression Rating (HDRS) total score, the proportion of participants achieving response (≥50% reduction in HDRS score at baseline) and the proportion of participants achieving remission (HDRS ≤12). The score ranges from 0-53 where a higher score is a worse outcome.
Edinburgh Postnatal Depression Scale | 8 weeks
  The mean change in scores of Edinburgh Postnatal Depression Scale. The scores range from 0 to 30 with 30 indicating more depression symptoms.
Generalized Anxiety Disorder 7-item scale | 8 weeks
  The mean change in scores of Generalized Anxiety Disorder 7-item scale. The scores range from 0 to 21. A higher generalized anxiety score indicates higher anxiety and indicating a worse outcome.
Young Mania Rating Scale | 8 weeks
  The mean change in scores of Young Mania Rating Scale. The YMRS is a rating scale used to evaluate manic symptoms at baseline and over time in individuals with mania. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. These four items are given twice the weight of the others. The score ranges from 0 to 60 where 60 indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Verinder Sharma, MB, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Parkwood Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There will be no sharing plan needed because no individual participant data (IPD) will be available to other researchers.